CLINICAL TRIAL: NCT01244061
Title: A Phase 4 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating The Efficacy And Safety Of Re-Treatment With Varenicline In Subjects Who Are Currently Smoking, And Who Have Previously Taken Varenicline
Brief Title: A Multi-National Study To Assess How Effective And Safe The Smoking Cessation Medicine Varenicline Is In Smokers Who Have Already Tried Varenicline In The Past As A Prescription Medicine From Their Usual Healthcare Provider
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051139
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline 1mg twice daily
  Arms: Varenicline
Drug: Placebo — Matched placebo twice daily
  Arms: Placebo

SUMMARY:
The main purpose of this study is to compare the effectiveness and safety of the re-treatment of smokers with varenicline with placebo for smoking cessation during the last 4 weeks of a 12 week course of treatment. The study will also assess whether smokers remain abstinent at Week 24 (12 weeks after the end of treatment) and Week 52 (40 weeks after the end of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Smokers aged 18 years or above and wanting to stop smoking
* Smokers who have smoked an average of at least 10 cigarettes per day over the last 4 weeks
* Smokers who have tried before to stop smoking at least once with varenicline, and who took varenicline for at least 2 weeks
* The last attempt to stop smoking must be at least 3 months before entering the study

Exclusion Criteria:

* Individuals who have not tolerated varenicline well previously, or who have a current or prior medical or psychiatric history that would make entry into the trial inadvisable
* Individuals who have previously participated in clinical trials of varenicline
* Individuals who have been participating in another smoking cessation trial within the last 3 months, or other drug trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (8):
  - Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - University of California Los Angeles David Geffen School of Medicine, Los Angeles, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - The University of Maryland, College Park, Maryland
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Oregon Health and Science University, Portland, Oregon
  - Clinical Research Associates, Inc., Nashville, Tennessee
- Australia (4):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - AusTrials Australia, Sherwood, Queensland
  - Emeritus Research, Malvern, Victoria
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Afdeling Pneumologie, Edegem
  - Universitaire Ziekenhuizen Leuven/Pneumologie, Leuven
  - Centre Hospitalier Universitaire de Liege, Liège
  - Cliniques Universitaires U.C.L. de Mont-Godinne/Laboratoire, Yvoir
- Canada (4):
  - Office of Dr. Ronald Collette, Burnaby, British Columbia
  - White Hills Medical Clinic, St. John's, Newfoundland and Labrador
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Clinique des maladies Lipidiques de Quebec, Québec, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Krajska nemocnice Liberec a.s., Plicni oddeleni, Liberec
  - Mestska nemocnice Ostrava, Plicni oddeleni, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (3):
  - CHU de la Cavale Blanche, Brest
  - CHU Côte de Nacre, Unité de Coordination de Tabacologie, Caen
  - Hopital Arnaud de Villeneuve, Montpellier
- Germany (5):
  - Universitaetsklinikum Goettingen Zentrum Innere Medizin Abteilung Kardiologie und Pneumologie, Göttingen, Germany
  - Klinische Forschung Berlin, Berlin
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Ludwig Maximilians-Universitaet Muenchen, München
  - FOCUS Clinical Drug Development GmbH, Neuss
- United Kingdom (5):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berks
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus Scotland Clinical Research Centre, Glasgow
  - Synexus, Merseyside Clinical Research Centre, Liverpool
  - William Harvey Research Institute,, London

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Gonzales D, Hajek P, Pliamm L, Nackaerts K, Tseng LJ, McRae TD, Treadow J. Retreatment with varenicline for smoking cessation in smokers who have previously taken varenicline: a randomized, placebo-controlled trial. Clin Pharmacol Ther. 2014 Sep;96(3):390-6. doi: 10.1038/clpt.2014.124. Epub 2014 Jun 9. PMID 24911368
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051139&StudyName=A%20Multi-National%20Study%20To%20Assess%20How%20Effective%20And%20Safe%20The%20Smoking%20Cessation%20Medicine%20Varenicline%20Is%20In%20Smokers%20Who%20Have%20Already%20Trie

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 4, randomized, double-blind, placebo-controlled, parallel group, 2-arm, multicenter study. A total of 498 participants were randomized into the study at 36 investigator sites.
Groups:
- Varenicline: Participants received 0.5 mg per day of varenicline on Days 1 to 3, 1.0 mg per day on Days 4 to 7, and 2.0 mg per day (1.0 mg twice daily, ie, 2 x 0.5 mg tablets in the morning and 2 x 0.5 mg tablets in the evening) from Weeks 1 to 12.
- Placebo: Participants received 1 tablet per day of placebo from Days 1 to 3, which was titrated up to 2 tablets per day from Days 4 to 7, and then to 4 tablets per day (2 tablets in the morning and 2 tablets in the evening) from Week 1 to Week 12.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 251 | 247
Completed | 169 | 144
Not Completed | 82 | 103
Not completed — Death | 1 | 0
Not completed — Did not meet entrance criteria | 1 | 0
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 34 | 30
Not completed — Withdrawal by Subject | 29 | 46
Not completed — Other | 8 | 19
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 5 | 2
Not completed — Randomized but not treated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 249 | 245 | 494
Age, Customized [Number; unit: number of participants]
  < 18 years | 0 | 0 | 0
  18-44 years | 94 | 94 | 188
  45-64 years | 135 | 139 | 274
  >= 65 years | 20 | 12 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 124 | 249
  Male | 124 | 121 | 245

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence Rate (CAR) From Week 9 Through Week 12
Description: The percentage of participants who, from Week 9 through Week 12, reported no smoking and no use of other nicotine-containing products since the last study visit/last contact (on the Nicotine Use Inventory) and who did not have carbon monoxide (CO)> 10ppm at any visits during this time frame.
Time Frame: Week 9 through Week 12
Population: The Full Analysis Set (FAS) included all participants as the primary participant population for efficacy analyses in this study and was defined as all participants who had received ≥1 dose, including partial doses, of randomized study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 249 | 245
Percentage of participants | 45.0 | 11.8
Statistical Analysis 1: Comparison: Varenicline vs Placebo; The study was conducted on a sample size to achieve at least 90% power for the treatment comparison in the primary efficacy endpoint assuming an odds ratio of 3.36 with a placebo abstinence rate of 12% and varenicline abstinence rate of 31%. The intent of the primary efficacy analysis was to evaluate the hypothesis that varenicline is superior to placebo for smoking cessation after 12 weeks of treatment; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — The statistical significance was declared for each hypothesis firstly for CAR Weeks 9-12, and then secondly for CAR Weeks 9-52 until a p-value > 0.05 was obtained, at which point the hypothesis would be declared to be not statistically significant; The analysis model included main effect of treatment and pooled center; Odds Ratio (OR) = 7.08, 95% CI 2-sided [4.34 to 11.55]

2. Secondary Outcome: CAR From Week 9 Through Week 52
Description: The percentage of participants who, from Week 9 through Week 52, reported no smoking (Weeks 9 through 52) and no use of other nicotine-containing products (Weeks 9 through 12), or no use of other tobacco products (Weeks 13 through 52), since the last study visit/last contact (on the Nicotine Use Inventory) and who did not have CO >10 ppm at any of these visits during this time frame.
Time Frame: Week 9 through Week 52
Population: The FAS included all participants as the primary participant population for efficacy analyses in this study and was defined as all participants who had received ≥1 dose, including partial doses, of randomized study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 249 | 245
Percentage of participants | 20.1 | 3.3
Statistical Analysis 1: Comparison: Varenicline vs Placebo; The sample size was sufficient to achieve 80% power for the treatment comparison in the key secondary end point for an odds ratio of 2.55 with a placebo abstinence rate of 6% and varenicline abstinence rate of 14%. The intent of the key secondary efficacy analysis was to evaluate the hypothesis that varenicline is superior to placebo for smoking cessation from Week 9 to the end of non-treatment follow up period at Week 52; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Statistical significance was declared for each hypothesis in the order above until a p-value >0.05 was obtained, at which point the hypothesis was declared to be not statistically significant; The analysis model included main effect of treatment and pooled center; Odds Ratio (OR) = 9.00, 95% CI 2-sided [3.97 to 20.41]

3. Secondary Outcome: CAR From Week 9 Through Week 24
Description: The percentage of participants who, from Week 9 through Week 24, reported no smoking (Weeks 9 through 24) and no use of other nicotine-containing products (Weeks 9 through 12), or no use of other tobacco products (Weeks 13 through 24), since the last study visit/last contact (on the Nicotine Use Inventory) and who did not have CO >10 ppm at any of these visits during this time frame.
Time Frame: Week 9 through Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 249 | 245
Percentage of participants | 28.9 | 7.8
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — The statistical test was two-sided and at a 0.05 level of significance. No adjustment was made for the analysis of multiple secondary endpoints; The analysis model included main effect of treatment and pooled center; Odds Ratio (OR) = 5.83, 95% CI 2-sided [3.25 to 10.44]

4. Secondary Outcome: 7-day Point Prevalence (PP) of Abstinence at Weeks 12, 24, and 52
Description: The secondary endpoint of 7-day point prevalence of smoking cessation was determined by evaluating a participant's cigarette smoking status, and other nicotine (and/or other tobacco) use, based on the "last 7 days" questions in the Nicotine Use Inventory. Additionally, a participant was not considered a responder if the expired CO was >10 ppm at the time point being summarized. Participants were considered responders independently at each visit.
Time Frame: Weeks 12, 24 and 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 249 | 245
Percentage of participants
  Week 12 | 53.0 | 14.7
  Week 24 | 32.9 | 15.5
  Week 52 | 28.9 | 12.2
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 12 assessment; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; The analysis model included main effect of treatment and pooled center; Odds Ratio (OR) = 7.85, 95% CI 2-sided [4.92 to 12.51]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Week 24 assessment; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; The analysis model included main effect of treatment and pooled center; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.86 to 4.64]
Statistical Analysis 3: Comparison: Varenicline vs Placebo; Week 52 assessment; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; The analysis model included main effect of treatment and pooled center; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.88 to 4.97]

ADVERSE EVENTS:
Time Frame: 2 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 7/249 | 4/245
Other Adverse Events (participants affected / at risk) | 145/249 | 70/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=249) | Placebo (N=245)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Allergy to chemicals (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=249) | Placebo (N=245)
Constipation (Gastrointestinal disorders) | 13 (13) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 0 (0)
Nausea (Gastrointestinal disorders) | 66 (87) | 22 (24)
Fatigue (General disorders) | 13 (14) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (19) | 17 (17)
Upper respiratory tract infection (Infections and infestations) | 19 (21) | 17 (17)
Headache (Nervous system disorders) | 26 (34) | 24 (32)
Abnormal dreams (Psychiatric disorders) | 36 (39) | 0 (0)
Insomnia (Psychiatric disorders) | 17 (19) | 0 (0)
Sleep disorder (Psychiatric disorders) | 13 (17) | 0 (0)

LIMITATIONS AND CAVEATS:
One SAE, exposure via semen, was not included under the Adverse Events since this event was considered to be experienced by a non-study participant, who was the study participant's partner. This event was coded as nonserious in the safety database.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.